CLINICAL TRIAL: NCT01099176
Title: The Effects of 90-day Monotherapies With Atorvastatin, Fenofibrate and Combined Therapy With Atorvastatin and Fenofibrate on Lipid Profile, Fasting Plasma Glucose, Proinflammatory Cytokines and Adipokines
Brief Title: Effects of Hypolipemic Treatment on Adipokines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Ministry of Scientific Research and Information Technology, Poland (Other Government)
Responsible Party: Okopień Bogusław MD, PhD, Medical University of Silesia, Dept. of Pharmacology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Ministry of Science
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2006-03

CONDITIONS: Hyperlipidemia; Impaired Fasting Glycemia
Keywords: hyperlipidemia; impaired fasting glycemia; adipokines; atorvastatin; fenofibrate
MeSH Terms: conditions — Hyperlipidemias | interventions — Psychotherapy, Multiple

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Atorvastatin (Experimental): 10mg of Atorvastatin
  Interventions: Drug: To compare monotherapies and combined therapy with each other
- Fenofibrate (Experimental): 267mg of Fenofibrate
  Interventions: Drug: To compare monotherapies and combined therapy with each other
- Fenofibrate and atorvastatin (Experimental): 10mg of Atorvastatin and 267mg of fenofibrate
  Interventions: Drug: To compare monotherapies and combined therapy with each other
- Therapeutic Lifestyle Change (Placebo Comparator): Placebo and Therapeutic Lifestyle Change
  Interventions: Drug: To compare monotherapies and combined therapy with each other

INTERVENTIONS:
Drug: To compare monotherapies and combined therapy with each other — Each patient received two tablets per day. Time interval between pills - 12 hours.
  In monotherapies patients received one active tablet and one placebo, in combined treatment both pills were active and in placebo group patients taken two placebo tablets

SUMMARY:
The study is planned to show whether monotherapies or combined hypolipemic therapy influence the fasting plasma glucose, serum adipokines (leptin, adiponectin, resistin) and proinflammatory cytokines (interleukin-6, TNF alpha) during 30 and 90 day course.

ELIGIBILITY:
Inclusion Criteria:

* Age (35-64yr)
* Primary hyperlipidemia (Total cholesterol >200mg/dl, Triglycerides >150mg/dl)
* Impaired fasting glycemia (glycemia 100-125mg/dl)
* For women:
* Menopause (>12 months)
* Post hysterectomy
* Mechanical contraception
* Obtained informed consent

Exclusion Criteria:

* Secondary hyperlipidemia
* Morbid obesity (BMI>40kg/m2)
* Alcohol or drug abuse
* Acute or chronic inflammation
* Congestive Heart Failure (NYHA III or IV)
* Unstable Ischaemic Heart Disease
* Moderate or severe hypertension
* Cancer in less than 5 years
* Chronic kidney disease (stage III-V)
* Liver failure
* Diabetes
* Oral contraception
* Not compliant patient
* Laboratory results:
* alanine transferase (>3xULN)
* creatine kinase (>5xULN)
* haemoglobin (<10/dl)
* PLT (<100G/l)
* WBC (<3,5G/l or >10G/l)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Adipokines | Day 90
  Serum concentration of leptin, adiponectin and resistin on Day 90 of the treatment.

SECONDARY OUTCOMES:
Proinflammatory cytokines | Day 30
  Interleukin-6 and TNF alpha serum concentration on the Day 30 of the treatment
Adipokines | Day 30
  Serum concentration of leptin, adiponectin and resistin on Day 30 of the treatment.
Proinflammatory cytokines | Day 90
  Interleukin-6 and TNF alpha serum concentration on the Day 90 of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacology, Katowice, Silesian Voivodeship, Poland